CLINICAL TRIAL: NCT01896115
Title: Current Steering to Optimize Deep Brain Stimulation
Brief Title: CUSTOM-DBS: Current Steering to Optimize Deep Brain Stimulation
Acronym: CUSTOM-DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: A4009; CDM00060272 (Other: BSC Protocol Number)
Record Dates: First submitted 2013-06-24; First posted 2013-07-11 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Parkinson's Disease
Keywords: Stimulation, implantable pulse generator, deep brain stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Short PW (Experimental): Patients with a Vercise DBS system programmed to 30 microseconds pulse width
  Interventions: Device: Vercise DBS settings
- Conventional PW (Experimental): Patients with a Vercise DBS system programmed to 60 microseconds pulse width
  Interventions: Device: Vercise DBS settings
- Ventral current steering (Experimental): Patients with a Vercise DBS system programmed to steer current ventrally
  Interventions: Device: Vercise DBS settings
- Dorsal current steering (Experimental): Patients with a Vercise DBS system programmed to steer current dorsally.
  Interventions: Device: Vercise DBS settings

INTERVENTIONS:
Device: Vercise DBS settings — Deep brain stimulation set at short pulse width and monopolar stimulation using current steering

SUMMARY:
The objective of the study is to compare different deep brain stimulation (DBS) settings using the commercially approved Boston Scientific Neuromodulation Vercise system.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, double-blind, randomized controlled trial.

This study will compare various program settings for the bilateral stimulation of the STN using the BSC implantable Vercise™ DBS System for the treatment of levodopa-responsive, moderate to severe idiopathic PD.

ELIGIBILITY:
Inclusion Criteria:

* Implanted bilaterally in STN with a Vercise DBS system for Parkinson's disease for at least three months with programming optimized according to standard of care.
* UPDRS subset III score of ≥30 in the in the pre-operative meds off state.
* DBS must improve PD symptoms by ≥30% in the meds off state, as measured by UPDRS subset III score.
* Medical and mental fitness to comply with programming visit and study related procedures.
* Able to understand the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed.
* Off symptom rigidity score of ≥2 in the evaluated arm as determined by the UPDRS-III.

Exclusion Criteria:

* Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, including any terminal illness with survival <12 months.
* Resting and/or action tremor score of ≥3 on the evaluated side as determined by the UPDRS-III in pre-operative meds off condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Neuromodulation Corporation
Locations (10):
- Boston Scientific Clinical Research Information toll free number, Valencia, California, United States
- A.o. LKH Univ.-Kliniken Innsbruck, Innsbruck, Austria
- Germany (5):
  - University Berlin, Charite Virchow, Berlin
  - Uniklinik Köln, Cologne
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - Universitatsklinikum Campus Kiel, Kiel
  - Universitaetsklinikum Wuerzburg, Würzburg
- Osp. S. Maria Della Misericordia, Udine, Italy
- United Kingdom (2):
  - Southmead Hospital Bristol, Bristol
  - Charing Cross Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects in Phase 1 received all Phase 1 treatments (Short PW, Conventional PW, Dorsal Steering, and Ventral Steering), so treatments are described as milestones below. The remaining 24 patients were assessed in Phase 2 for secondary/exploratory endpoints comparing single contact stimulation vs. current steering.
Pre-assignment Details: Interim analysis showed 16 patients to be a sufficient sample size for primary endpoints.
Groups:
- All Arms (Phase 1): Patients with a Vercise DBS system programmed to 30 microseconds pulse width
  Patients with a Vercise DBS system programmed to 60 microseconds pulse width
  Patients with a Vercise DBS system programmed to steer current ventrally
  Patients with a Vercise DBS system programmed to steer current dorsally.
- All Arms (Phase 2): Patients with a Vercise DBS system programmed to 30 microseconds pulse width
  Patients with a Vercise DBS system programmed to 60 microseconds pulse width
  Patients with a Vercise DBS system programmed to steer current
  Patients with a Vercise DBS system programmed to single contact stimulation
Period: Overall Study
Arm/Group | All Arms (Phase 1) | All Arms (Phase 2)
Started | 16 | 24
Phase 1 Short PW | 15 | 0
Phase 1 Conventional PW | 15 | 0
Phase 1 Dorsal Steering | 15 | 0
Phase 1 Ventral Steering | 15 | 0
Phase 2 Single Contact | 0 | 24
Phase 2 Steering | 0 | 24
Completed | 15 | 24
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Arms (Phase 1): Patients with a Vercise DBS system programmed to 30 microseconds pulse width
- All Arms (Phase 2): Patients with a Vercise DBS system programmed to 60 microseconds pulse width
- Total: Total of all reporting groups
Arm/Group | All Arms (Phase 1) | All Arms (Phase 2) | Total
Number analyzed (Participants) | 15 | 24 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (7.73) | 54.0 (8.43) | 56.5 (8.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Window
Description: The therapeutic window refers to the range of stimulus amplitudes that provide a therapeutic effect without side effects. In other words, it is the amplitude difference between the first stimulation-induced side effect threshold (e.g., eye deviation, muscle contraction, and speech) and full rigidity control threshold at 60 µs and 30 µs pulse width DBS settings.
Time Frame: Day 1 programming visit
Population: Therapeutic window for current steering settings was not a primary outcome measure but is described later as an "Other" outcome measure.
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Short PW | Conventional PW
Number analyzed (Participants) | 15 | 15
mA | 3.81 (2.78) | 2.32 (1.45)

2. Primary Outcome: Unified Parkinson's Disease Rating Scale III
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) has four sections (I-IV) that ask patients to rate aspects of their mental state including mood (I), aspects of daily activities (II), aspects of motor function (III), and complications of treatment (IV). Here, we ask subjects to rate their motor function (UPDRS III) following interventions with 30 µs and 60 µs pulse width DBS settings.
  The UPDRS III scale has 14 categories including speech, facial expression, tremor at rest, action tremor, rigidity, finger tapping ability, ability to open and close hands, ability to rapidly alternate hand movements, leg agility, ability to rise from a chair, posture, gait, response to postural displacement (e.g., push), and bradykinesia. Patients rate each of these categories from 0 to 4, with 0 being normal function and 4 being the worst. Categories assessing appendages are rated for both left and right sides, allowing a maximum score (worst outcome) of 108.
Time Frame: Day 1 programming visit
Population: All subjects were analyzed at both pulse widths. Primary outcomes were only intended to be assessed for different pulse widths and not current steering.
Measure: Mean (Standard Deviation); unit: UPDRS III score
Arm/Group | Short PW | Conventional PW
Number analyzed (Participants) | 15 | 15
UPDRS III score | 31.9 (11.55) | 31.3 (10.99)

3. Secondary Outcome: Side Effect Thresholds - Single Contact vs. Steering
Description: This endpoint determined how much current (mA) could be applied before side effects appeared when using 60 microsecond pulse widths. Values were obtained for when current was delivered through a single contact or divided between two contacts (steering).
Time Frame: Day 1 programming visit
Population: The 24 patients reported here are a separate population from the 16 patients who were enrolled for primary endpoint analysis (40 total patients).
Measure: Mean (Standard Deviation); unit: mA
Groups:
- Single Contact; Current Steering: All 24 patients analyzed for secondary endpoints received both single contact stimulation and current steering stimulation.
Arm/Group | Single Contact | Current Steering
Number analyzed (Participants) | 24 | 24
mA | 5.3 (2.3) | 5.2 (1.8)

4. Secondary Outcome: Resting Tremor Severity - Single Contact vs. Steering
Description: Resting tremor was measured by a motion sensor system (Kinesia System) while either using a single contact or steering current between two contacts. Stimulation was at amplitudes defined as the therapeutic threshold for rigidity. The Kinesia System was worn by patients to measure motion parameters including linear acceleration and angular velocity during different tasks, then provided an output score on a scale of 0 (no symptoms) to 4 (severe symptoms).
Time Frame: Day 1 programming visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Contact | Current Steering
Number analyzed (Participants) | 24 | 24
units on a scale | 0.2 (0.6) | 0.2 (0.6)

5. Secondary Outcome: Finger Tapping Amplitude - Single Contact vs. Steering
Description: Severity of finger-tapping bradykinesia was measured by a motion sensor system (Kinesia System) when either using a single contact or steering current between two contacts. Stimulation was at amplitudes defined as the therapeutic threshold for rigidity. The Kinesia System was worn by patients to measure motion parameters including linear acceleration and angular velocity during different tasks, then provided an output score on a scale of 0 (no symptoms) to 4 (severe symptoms).
Time Frame: Day 1 programming visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Contact | Current Steering
Number analyzed (Participants) | 24 | 24
units on a scale | 2.2 (0.9) | 2.3 (0.7)

6. Other Pre Specified Outcome: Dorsal-Ventral Current Steering Therapeutic Window
Description: The therapeutic window refers to the range of stimulus amplitudes that provide a therapeutic effect without side effects. In other words, this measure reports the stimulus amplitude difference between the full rigidity control threshold and the first stimulation induced side effect threshold at current steering settings (current divided 50% between adjacent electrodes).
Time Frame: Day 1 programming visit
Population: The therapeutic window of short pulse widths vs. conventional pulse widths was a primary outcome measure and is reported as such in another section of this report.
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Ventral Current Steering | Dorsal Current Steering
Number analyzed (Participants) | 15 | 15
mA | 2.05 (1.82) | 2.56 (2.76)

7. Other Pre Specified Outcome: Resting Tremor Severity - Pulse Width and Dorsal-Ventral Steering
Description: Resting tremor was measured by a motion sensor system (Kinesia System) at 60 µs, 30 µs, and current steering settings, at amplitudes defined as the therapeutic threshold for rigidity. The Kinesia System was worn by patients to measure motion parameters including linear acceleration and angular velocity during different tasks, then provided an output score on a scale of 0 (no symptoms) to 4 (severe symptoms).
Time Frame: Day 1 programming Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Short PW | Conventional PW | Ventral Current Steering | Dorsal Current Steering
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale | 0.25 (0.63) | 0.34 (0.71) | 0.13 (0.34) | 0.30 (0.62)

8. Other Pre Specified Outcome: Finger Tapping Amplitude - Pulse Width and Dorsal-Ventral Steering
Description: Severity of finger-tapping bradykinesia was measured by a motion sensor system (Kinesia System) at 60 µs, 30 µs, and dorsal and ventral current steering settings. Stimulation was at amplitudes defined as the therapeutic threshold for rigidity. The Kinesia System was worn by patients to measure motion parameters including linear acceleration and angular velocity during different tasks, then provided an output score on a scale of 0 (no symptoms) to 4 (severe symptoms).
Time Frame: Day 1 programming visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Short PW | Conventional PW | Ventral Current Steering | Dorsal Current Steering
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale | 2.16 (0.74) | 2.20 (0.63) | 2.17 (0.77) | 2.16 (0.73)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Patients in this study only had 1 visit. Adverse event data were not collected for Phase 2.
Groups:
- All Arms: Patients with a Vercise DBS system programmed to 4 different settings including:
  1. Short pulse widths (30 microseconds)
  2. Conventional pulse widths (60 microseconds)
  3. Steering current ventrally
  4. Steering current dorsally
Arm/Group | All Arms
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No